CLINICAL TRIAL: NCT03859141
Title: Open Phase I and Randomized, Double-blind, Controlled Phase III Clinical Trial to Evaluate the Safety and Immunogenicity of Quadrivalent Influenza Vaccine in Healthy Subjects Aged 6-35 Months
Brief Title: Clinical Trial to Evaluate the Safety and Immunogenicity of Quadrivalent Influenza Vaccine (7.5μg/0.25ml)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-QINF-3002
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Seasonal Influenza
Keywords: Influenza Vaccine; Quadrivalent; Trivalent; Children
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: The phase Ⅰ clinical trial was a single arm.The phase Ⅲ was 3 parallel arms.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group-phase Ⅰ (Experimental): Quadrivalent influenza vaccine
  Interventions: Biological: Quadrivalent influenza vaccine
- Experimental group-phase Ⅲ (Experimental): Quadrivalent influenza vaccine
  Interventions: Biological: Quadrivalent influenza vaccine
- Control group 1-phase Ⅲ (Active Comparator): Trivalent influenza vaccine (contains B/Victoria strain)
  Interventions: Biological: Trivalent influenza vaccine (contains B/Victoria strain)
- Control group 2-phase Ⅲ (Active Comparator): Trivalent influenza vaccine (contains B/Yamagata strain)
  Interventions: Biological: Trivalent influenza vaccine (contains B/Yamagata strain)

INTERVENTIONS:
Biological: Quadrivalent influenza vaccine — One dose of quadrivalent influenza vaccine: 0.25 ml per dose containing 7.5μg antigen.
  Arms: Experimental group-phase Ⅰ
Biological: Quadrivalent influenza vaccine — One dose of quadrivalent influenza vaccine: 0.25 ml per dose containing 7.5μg antigen.
  Arms: Experimental group-phase Ⅲ
Biological: Trivalent influenza vaccine (contains B/Victoria strain) — One dose of trivalent influenza vaccine (contains B/Victoria strain): 0.25 ml per dose containing 7.5μg antigen.
  Arms: Control group 1-phase Ⅲ
Biological: Trivalent influenza vaccine (contains B/Yamagata strain) — One dose of trivalent influenza vaccine (contains B/Yamagata strain): 0.25 ml per dose containing 7.5μg antigen.
  Arms: Control group 2-phase Ⅲ

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of quadrivalent influenza vaccine in healthy children aged 6-35 months.

DETAILED DESCRIPTION:
The study includes open-labelled phase I and randomized, double-blind, controlled phase III clinical trial. In the phase I, 20 healthy Chinese children aged 6-35 months were administered with two doses of QIV (7.5μg/0.25ml). In the phase Ⅲ clinical trial, 2320 children were assigned to QIV group, TIV (B/Victoria) group and TIV (B/Yamagata) group in a 2:1:1 ratio. All vaccines were manufactured by Sinovac Biotech Co., Ltd.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer between 6 - 35 months old; Term birth; Birth weight >2500g;
* Proven legal identity;
* Written consent of the guardian(s) of the volunteer;

Exclusion Criteria:

* Received seasonal influenza vaccine in the current year;
* Suffering from seasonal influenza in the past 6 moths;
* Axillaty temperature > 37.0 °C;
* History of allergy to any vaccine or vaccine ingredient;
* History of serious adverse reaction(s) to vaccination, such as urticaria, difficulty in breathing, angioneurotic edema, abdominal pain, etc;
* Autoimmune disease or immunodeficiency;
* Congenital malformation, developmental disorders;
* Severe malnutrition;
* Diagnosed coagulation function abnormal (e.g., coagulation factor deficiency, coagulation disorder, or platelet abnormalities) , or obvious bruising or coagulation disorders;
* History of epilepsy (except febrile seizures occurred < 2 years of age or pure epilepsy occurred within the past 3 years that does not need treatment)
* Chronic diseases (e.g., viral hepatitis, tuberculosis, diabetes, blood diseases, or neurological disorders)
* Acute disease or acute stage of chronic disease;
* Receipt of any of the following products:

  1. Any subunit vaccine or inactivated vaccine (e.g., pneumococcal vaccine) or treatment of allergy within 14 days prior to study entry;
  2. Any live attenuated vaccine within 30 days prior to study entry;
  3. Any other investigational medicine(s) or vaccine within 30 days prior to study entry;
  4. Blood product within 3 months prior to study entry;
  5. Any immunosuppressant, cytotoxic medicine, or inhaled corticosteroids (except corticosteroid spray for treatment of allergic rhinitis or corticosteroid treatment on surface for acute non-complicated dermatitis) within 6 month prior to study entry;
* Participate or will participate in other clinical trial(s) during this study;
* Based on the judgment of investigator(s) or the Ethic Committee, there was any condition indicating that the subject should be excluded;

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2340 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
The lower limit of 95% confidence intervals (95%CI) of geometric mean titer (GMT) ratio (experimental group/control group) of hemagglutination inhibition (HI) antibody titer≥2/3. | 28 days after two doses immunization
  Immunogenicity index, One of the standard to evaluate the experimental vaccine is non-inferior to the control vaccines.
The lower limit of 95% CI of the seroconversion rate difference (experimental group-control group)≥-10%. | 28 days after two doses immunization
  Immunogenicity index, Another standard to evaluate the experimental vaccine is non-inferior to the control vaccines.

SECONDARY OUTCOMES:
The lower limit of 95%CI of the ratio of GMT (experimental group/control group) >1.5. | 28 days after two doses immunization
  Immunogenicity index, One of the standard to evaluate the experimental vaccine is superior to the control vaccines for specific antigen type.
The lower limit of 95% CI of the difference of HI antibody seroconversion rate (experimental group-control group)>10% | 28 days after two doses immunization
  Immunogenicity index, Another standard to evaluate the experimental vaccine is superior to the control vaccines for specific antigen type.
The lower limit of 95% CI of seroconversion rate for each HI antibody after two doses immunization≥40%. | 28 days after two doses immunization
  Immunogenicity index
The seroprotective rate (HI antibody titer≥1:40) of each HI antibody after two doses immunization≥70%. | 28 days after two doses immunization
  Immunogenicity index
The geometric mean increase (GMI) of each HI antibody after two doses immunization >2.5. | 28 days after two doses immunization
  Immunogenicity index
The lower limit of 95%CI of the ratio of GMT(experimental group/control group)≥2/3, in the subjects whose pre-immune HI antibody titer<1:40 | 28 days after two doses immunization
  Immunogenicity index
The lower limit of 95% CI of the difference of HI antibody seroconversion rate (experimental group-control group)≥-10%, in the subjects whose pre-immune HI antibody titer<1:40. | 28 days after two doses immunization
  Immunogenicity index
The incidence of the solicited local and general adverse reactions 0-7 days after each immunization. | 0-7 days
  Safety index, The adverse reactions refers to the adverse events which were considered related to the vaccination.
The incidence of the unsolicited adverse events 0-28 days after each immunization | 0-28 days after each dose immunization
  Safety Index
The incidence of the serious adverse events within 7 months after the first immunization. | Within 7 months after the first dose immunization
  Safety Index

CONTACTS AND LOCATIONS:
Overall Officials: Yuemei Hu, Bachelor, Principal Investigator — Jiangsu Provincial Center for Disease Prevention and Control
Locations (2):
- China (2):
  - Guanyun Center for Disease Prevention and Control, Lianyungang, Jiangsu
  - Pizhou Center for Disease Prevention and Control, Pizhou, Jiangsu

REFERENCES:
- [Derived] Hu Y, Shao M, Hu Y, Liang Q, Jia N, Chu K, Xu L, Li J, Li C, Zhu F. Immunogenicity and safety of an inactivated quadrivalent influenza vaccine: a randomized, double-blind, controlled phase III clinical trial in children aged 6-35 months in China. Hum Vaccin Immunother. 2020 Jul 2;16(7):1691-1698. doi: 10.1080/21645515.2020.1721994. Epub 2020 Apr 29. PMID 32347785